CLINICAL TRIAL: NCT06734455
Title: Robot-Assisted Laparoscopic Pyeloplasty in Children Younger Than 5 Years Old
Brief Title: Robot-Assisted Pyeloplasty in Young Children
Acronym: PYEROB
Status: Completed | Type: Observational
Sponsor: Destinval Christelle (Other)
Responsible Party: Sponsor-Investigator, Destinval Christelle, M.D., University Hospital, Clermont-Ferrand
Organization: University Hospital, Clermont-Ferrand (Other)
Other Study IDs: M24DC1107; NCT05858658 (obsolete NCT alias)
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2022-12

CONDITIONS: Ureterohydronephrosis; Ureter Obstruction; Child, Only
Keywords: Robot-Assisted Pyeloplasty; Child; Retrospective Study
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Robot-Assisted Pyeloplasty — Pyeloplasty in Children using robotic surgery

SUMMARY:
The goal of this retrospective study is to analyse the outcomes of Robot-Assisted Pyeloplasty in participants younger than 5 years old:

* indication criteria
* clinical symptoms
* operating time
* length of stay
* complications
* follow-up

DETAILED DESCRIPTION:
Outcomes of Robot-Assisted Pyeloplasty in participants younger than 5 years old and comparison with the outcomes in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 5 years old, who underwent primary robotic pyeloplasty, was launched between January 2014 and December 2022

Exclusion Criteria:

* Patients older than 5 years old, who underwent primary robotic pyeloplasty, was launched between January 2014 and December 2022

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients younger than 5 years old, with pyeloureteric syndrome, who underwent primary robotic pyeloplasty
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Presence of ureterohydronephrosis | Before surgery
  Ureterohydronephrosis represents the augmentation of the diameter of the ureter (more than 10 millimeters) and the renal pelvis (more than 30 millimeters), which can be measured on imaging such as abdominal ultrasound, CT scan, or MRI. Whenever the ureter and the renal pelvis meet these criteria on preoperative imaging, the patient will be labeled as having ureterohydronephrosis.
Presence of abdominal pain | Before surgery
  Flank pain (pain in the upper abdomen or back)
Presence of urinary calculi | Before surgery
  Urinary calculi can be diagnosed on an abdominal X-Ray, an abdominal Ultrasound or an abdominal CT scan
Presence of abnormal nuclear renal scans | Before surgery
  Nuclear renal scans are abnormal when there is a difference of filtration of more than 40% between the kidneys
Presence of urinary tract infection | Before surgery
  Urinary tract infection associated with ureteropelvic junction

SECONDARY OUTCOMES:
Postoperative pain | After surgery and before discharge home, up to 20 days
  The numeric rating scale (NRS) is a pain screening tool commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and ten meaning "the worst pain imaginable."
Postoperative complications | Through study completion, an average of 2 years
  Pyelonephritis
Operation time | During surgery
  anesthetic and operating time
Hospitalization length | From admission to discharge home, up to 20 days
  Hospitalization length

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization the investigators won't share individual participant data

REFERENCES:
- [Background] Esposito C, Cerulo M, Lepore B, Coppola V, D'Auria D, Esposito G, Carulli R, Del Conte F, Escolino M. Robotic-assisted pyeloplasty in children: a systematic review of the literature. J Robot Surg. 2023 Aug;17(4):1239-1246. doi: 10.1007/s11701-023-01559-1. Epub 2023 Mar 13. PMID 36913057